CLINICAL TRIAL: NCT01616290
Title: Open-Label, Dose-Escalation, Pilot Study of PRT-201 Administered Following Angioplasty in Patients With Peripheral Artery Disease in the Lower Extremity
Brief Title: Pilot Study of PRT-201 Following Angioplasty in Patients With Peripheral Artery Disease (PAD)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Proteon Therapeutics (Industry)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRT-201-103
Record Dates: First submitted 2012-06-06; First posted 2012-06-11 (Estimated); Last update posted 2015-08-11 (Estimated); Status verified 2015-08

CONDITIONS: Peripheral Artery Disease
Keywords: peripheral artery disease; PAD; claudication; angioplasty; percutaneous transluminal angioplasty; PTA; superficial femoral artery; SFA; popliteal artery; PA; PRT-201; restenosis; vonapanitase
MeSH Terms: conditions — Peripheral Arterial Disease; Intermittent Claudication | interventions — cholesterol-binding protein

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: PRT-201 — 0.03, 1, or 3 mg single adventitial administration

SUMMARY:
The purpose of this study is to determine if it is safe and feasible to apply PRT-201 to the adventitia of arteries following successful angioplasty (PTA).

ELIGIBILITY:
Inclusion Criteria:

1. Age of at least 18 years
2. Clinical diagnosis of PAD, secondary to atherosclerosis affecting a lower limb
3. Rutherford classification 2-4 (moderate claudication to ischemic rest pain)
4. ABI <0.90 at rest or with exercise, or a toe-brachial index <0.70, or radiographic evidence of PAD that correlates with clinical symptoms
5. De novo lesion, not previously treated by angioplasty or atherectomy
6. Greater than 70% stenosis of the SFA or PA, target lesion length of 10 cm or less, and at least one patent runoff vessel. Short segment occlusions (<10 cm) are acceptable
7. If female and of childbearing potential (premenopausal and not surgically sterile) must have a negative pregnancy test at the screening visit and be willing to use contraception from the time of the screening visit to 1 week following study drug administration. Acceptable methods of birth control include abstinence, barrier methods with spermicide, implants, injectables, oral contraceptives, intra-uterine device, or a vasectomized partner
8. Ability to understand and comply with the requirements of the entire study and communicate with the study team
9. Ability to provide written informed consent using a document that has been approved by the required institutional review board

Exclusion Criteria:

1. Previous treatment with PRT-201
2. Patients in whom arterial insufficiency in the lower extremity is the result of an immunologic or inflammatory non-atherosclerotic disorder (e.g. Buerger's disease, vasculitis)
3. Current severe critical limb ischemia defined as ulceration or gangrene
4. Planned atherectomy of the arteries of the index leg
5. Prior or planned stenting of the target lesion
6. Prior bypass surgery to the target SFA or PA
7. Severe concentric medial calcification of the target lesion thought to interfere with drug delivery to the adventitia that is defined subjectively by the Investigator based on fluoroscopic appearance.
8. History of metastatic cancer
9. Presence of aortic or peripheral artery aneurysm
10. Platelet count <130K, hematocrit <30%, bilirubin or ALT >3.0 times the upper limit of normal
11. Pregnancy, lactation or plans to become pregnant during the course of the study
12. Presence of any significant medical condition that might significantly confound the collection of safety and efficacy data in this study
13. Treatment with any investigational drug within the previous 30 days or investigational antibody therapy within 90 days prior to signing informed consent
14. Known allergy to contrast media

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-10; Primary Completion 2014-06 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Clinical Safety | 12 months following PTA and study drug administration
  Safety evaluations will be based on adverse events, physical examinations, ultrasounds, vital signs, and clinical laboratory results. Events of interest (EOI) include: acute occlusion, vessel dissection, vessel rupture, aneurysm, pseudoaneurysm, target lesion revascularization, limb amputation, and death.

SECONDARY OUTCOMES:
Technical success of adventitial administration of PRT-201 | Immediately following study drug administration
  Technical success of study drug administration will be assessed by the extent of circumferential and longitudinal coverage of the artery by the study drug. A standardized scale will be used to grade the pattern of distribution for each patient.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher D Owens, M.D., M.Sc, Principal Investigator — San Francisco VA Medical Center
Locations (2):
- United States (2):
  - San Francisco VA Medical Center, San Francisco, California
  - University of California, San Francisco Medical Center, San Francisco, California